CLINICAL TRIAL: NCT05073289
Title: EXAMINATION OF THE EFFECT OF" SANDPLAY ACTIVITY " ON ANXIETY AND WELL-BEING IN PATIENTS IN A PSYCHIATRIC CLINIC
Brief Title: Sandplay Activity in Psychiatry Clinic (SAPC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sema Soysal, Investigator, Akdeniz University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: SSoysal
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Sandplay Therapy; Anxiety
Keywords: anxiety, well-being, sandplay, psychiatric nursing, psychiatric care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Control Experimental Research
Who Masked: Participant
Masking Description: Patients with a diagnosis of mental disorder in the psychiatry clinic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAPC (Experimental): SAPC is a acronmy that defines Sandplay activity in psychiatry clinic
  Interventions: Behavioral: Sandplay activity
- Control Group (Active Comparator)
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: Sandplay activity — The sandplay in psychiatric care, with a creative and fun approach, makes it easier for patients to verbally express their personal life stories and feelings in a safe environment, individually or as a group.
  Arms: SAPC
Other: Routine Care — Routine care is the care given to the control group by the nurse to the patients in the psychiatry clinic.
  Arms: Control Group

SUMMARY:
This research was conducted to examine the effect of sandplay activity on anxiety and well-being levels in patients in psychiatric clinics.

The research was carried out in Isparta Süleyman Demirel University Psychiatric Clinic as a single-blind randomized controlled experimental study in the pre-test, final-test order between 2020-2021. Ethical permission was obtained from the Clinical Research Ethics Committee and application permission from the institution for pre-research. 63 patients (intervention-32 and control-31) selected by block randomization method formed the universe of the study. No intervention was applied to the control group. A preliminary test and a final test were performed two days apart, one hour apart on the first and fourth days. Two sessions of sandplay activity were applied to the intervention group with a decongest of two days, and each session was pre-tested. The data was collected using "The Personal Information Form", "The Spielberger Status Anxiety" inventory, and "Well-Being Star Scale" and also data showed normal distribution. In statistical analysis, T-Test, Chi-Square Test, pearson correlation test was used dependent and independent groups.

For the purpose of the research, the hypotheses of the research are as follows::

1. Hypothesis (H1): after intervention, anxiety levels of patients who underwent sandplay activity (in a psychiatric clinic) are lower than in the control grouproup
2. Hypothesis (H1): after intervention the level of well-being of patients undergoing sand play activity (in a psychiatric clinic) is higher than that of the control group.
3. Hypothesis (H1): there is a negative correlation between the level of anxiety and the level of well-being in psychiatric clinics who sandplay activity is practiced and not practiced.

This research is Turkish language.

ELIGIBILITY:
Inclusion Criteria Being over 18 years old, Volunteering to participate, Not having a defect in the ability to evaluate and reason the truth, Not having hearing, understanding, and speaking problems, Not have a physical disability

Exclusion Criteria from Research To be involved in another study on a similar experimental subject Being on the first day of hospitalization and on the day of discharge

Removing Criteria State their willingness to leave the research voluntarily Transfer to another place and/or unscheduled early discharge

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
"Spielberger Status Anxiety Inventory" | 4 days changes after the first interview
"Well-being Star Scale" | 4 days changes after the first interview

CONTACTS AND LOCATIONS:
Locations (1):
- Sema Soysal, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No